CLINICAL TRIAL: NCT04413006
Title: A Self-compassion Group-based Treatment for Chronic Pain Via Video Conferencing During the COVID-19 Pandemic: Feasibility Study for a Potential New Mode of Treatment Delivery
Brief Title: Self-compassion for Chronic Pain Virtual Group Treatment Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sccpvgtbsas2020
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain
Keywords: Virtual treatment; Group Treatment; Self-Compassion
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants who will receive the 6-session Group-Based Virtual Self-Compassion for Chronic Pain treatment
  Interventions: Behavioral: Self-Compassion for Chronic Pain Virtual Group Treatment Program

INTERVENTIONS:
Behavioral: Self-Compassion for Chronic Pain Virtual Group Treatment Program — 6-session group via video-conferencing for informational and experiential exercises to increase self-compassion in individuals with chronic pain

SUMMARY:
As a result of COVID-19 and measures taken by the Canadian Government to reduce the transmission of the virus, in-person psychology services have been suspended. Psychology services are now being conducted via video conferencing. The purpose of the current project is to pilot-test a 6-week Self Compassion Treatment for Chronic Pain delivered virtually, in order to understand its utility in the current environment. The treatment is to be delivered through a secure professional ZOOM licence. Objective 1 of the project is to assess the feasibility and acceptability of attending the treatment group through virtual participation. Objective 2 is to assess the effectiveness of the group treatment in improving self-compassion, mental health, relationship with pain, and quality of life.

DETAILED DESCRIPTION:
Participants will be adult psychology outpatients of one of the two tertiary care pain clinics in Winnipeg, or patients of one of the psychologists working in the Clinical Health Psychology Program, and who would normally have been invited to attend an in-person group-based intervention at the Health Sciences Centre.

Participants will complete a set of questionnaires that are standard in our clinic, and that will be accessed via the online survey platform, Survey Gizmo.

Participants will complete 6-weeks of the virtual Self-Compassion for Chronic Pain Treatment Group. Session 1: Participant introductions. Introduction of concepts: Self-Compassion (and how it differs from Self-Esteem, Self-Pity, or Self-Indulgence), rationale of self-compassion for chronic pain. Introductory experiential self-compassion exercises. Assignment of homework. Session 2: Check-in and homework review. Introduction to mindfulness and its applicability in self-compassion. Brief body scan and mindfulness of the breath exercises. ACT Matrix exercise. Additional experiential self-compassion exercises. Discussion of awareness of pleasant experiences. Assignment of homework (including awareness of pleasant experiences throughout the week). Session 3: Check-in and homework review. Self-Compassion in relationships and being present and compassionate in our relationships. Loving-kindness meditation. Additional experiential self-compassion exercises Assignment of homework. Session 4: Check-in and homework review. Self-Compassion in the face of difficulties. Working with difficult emotions (e.g., shame, guilt, anger, self-criticism) with self-compassion. Additional experiential self-compassion exercises. Assignment of homework. Session 5: Check-in and homework review. Self-care in chronic pain management. Cultivating gratitude, self-appreciation and savouring attitudes. Additional experiential self-compassion exercises. Assignment of homework. Session 6: Check-in and homework review. Compassionate body scan. Review of program. A look forward (strategies to maintain practices, prepare for setbacks and get back on track). Wrap-up.

Procedure. All participants who were scheduled to attend an in-person group-based therapy program will be contacted to invite them to participate in this new virtual group. They will be assured that their decision to participate (or to not participate) in this study will not impact their eligibility for participation in the next in-person group, when in-person groups resume. Additionally, current patients of pain psychologists in the Clinical Health Psychology Program will be invited to the new program at the discretion of the treating psychologist (this is in line with current practices). They will be informed that because they are participating in a new group, a novel delivery format, and a unique environment, the group program will be evaluated as part of a research study. If they agree to be part of the study verbally, they will be sent a link to the Consent form and baseline questionnaires through Survey Gizmo. Baseline questionnaires will be reviewed prior to beginning of the group, and all participants who score in the "severe" range on the PHQ-9 (i.e. a score of 20 or higher), or who score a "2 or higher" on item number 9 (Thoughts that you would be better off dead, or thoughts of hurting yourself in some way) will be contacted by telephone for further screening. They may then be offered individual distance therapy rather than the group-based therapy, as per Dr. Sabourin's assessment. All consented participants will be contacted by one of the two therapists (Ms. Amanda Shamblaw, Psychology Resident or Dr. Brigitte Sabourin, PhD, CPsych) prior to beginning the group in order to test out the connection and problem-solve any difficulties. They will also be given some preliminary instructions regarding attending a video-based appointment, as per the Clinical Health Psychology Program's guidelines. These include a 2-part verification of patient identification (date of birth and Patient health identification number - PHIN), informing participants that "Despite our best efforts to ensure high level of privacy and secure technology, there is always a risk that the transmission be breached and accessed by unauthorized persons", "no sessions are recorded", "no personal information is shared with Zoom". They will then verbally consent to proceed. Participants will participate in the 6 weekly sessions in groups of 10-12 participants. At the beginning of each session, each participant will be in a virtual "waiting room", and either Ms. Shamblaw or Dr. Sabourin will confirm the participant's location and phone number prior to admitting them to the group. The location and phone numbers are collected in order to be able to reach participants if needed. They will complete measures post-treatment and at a 3-month follow-up using Survey Gizmo. Finally, following treatment, participants will have the option to participate in a semi-structured qualitative interview to discuss their impressions of the group, impressions of attending virtually, support they felt from other group members, and general group cohesion feedback. Participants will be informed that the interview is voluntary and will not affect their participation in the treatment group.

ELIGIBILITY:
Inclusion Criteria: Seeking services from a Chronic Pain Specialty Services (tertiary care multi-disciplinary clinic, or health psychologist). Having sufficient internet capacity to participate in the video conferences, and proficiency in speaking and understanding English -

Exclusion Criteria: severe depressive symptoms; acute suicidality

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change over time in Scores on the Self-Compassion Scale (SCS) | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the Self-Compassion Scale (SCS) (score range is 12-60 with increases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Change over time in Scores on the Pain Disability Index | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the Pain Disability Index (score range is 0-70 with decreases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)

SECONDARY OUTCOMES:
Change over time in Scores on the Chronic Pain Acceptance Questionnaire - 8 | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the on the Chronic Pain Acceptance Questionnaire - 8 (CPAQ-8) (score range is 0-48 with increases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Change over time in Scores on the Pain Catastrophizing Scale -6 | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the on the Pain Catastrophizing Scale-6 (PCS-6) (score range is 0-24 with decreases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Change over time in Scores on the Pain Self-Efficacy Questionnaire-4 | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in Scores on the Pain Self-Efficacy Questionnaire-4 (PSEQ-4) (score range is 0-24 with increases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Change over time in Pain Intensity | at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the Numeric Rating Scale (NRS) for pain (score range is 0-10 with decreases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Change over time in Depression Symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the Patient Health Questionnaire-9 (PHQ-9) (score range is 0-27 with decreases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Changes over time in Anxiety Symptoms as measured by the Generalized Anxiety Scale-7 | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the Generalized Anxiety Scale (GAD-7) (score range is 0-21 with decreases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Change over time in Quality of Life as measured by the PROMIS GLOBAL- 10 | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Change over time in scores on the Physical Health and Mental Health Quality of Life scores from the PROMIS GLOBAL-10 (score range is 7-35 with increases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)
Changes over time in Mindfulness | baseline, at treatment end (6-weeks after beginning treatment) and 3 months later
  Changes over time in score on the Mindfulness Attention and Awareness Scale (MAAS) (score range is 15-90 with increases in scores meaning better outcome). Change over time to be assessed via repeated measures Analysis of Variance (ANOVA)

OTHER OUTCOMES:
Client Satisfaction | post treatment (6 weeks after beginning the treatment)
  Scores on the Client Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Sabourin, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada